CLINICAL TRIAL: NCT04895345
Title: An Open, Single-arm, Single-center, Phase II Clinical Trial of TQB2450 in Combination With Intensity-modulated Radiotherapy in Patients With Inoperable Locally Recurrent Nasopharyngeal Carcinoma
Brief Title: A Study of TQB2450 in Combination With Intensity-modulated Radiotherapy in Patients With Inoperable Locally Recurrent Nasopharyngeal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2450-II-11
Record Dates: First submitted 2021-05-17; First posted 2021-05-20 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2450+Intensity modulated radiotherapy (Experimental): TQB2450 1200 mg administered intravenously (IV) on Day 1 of each 21-day；The total dose of radiotherapy should meet PTVnx: 60Gy/27Fr/2.22Gy, PTVnd: 60-64Gy/27Fr/2.22-2.37Gy, PTV1: 54Gy/27Fr/2.00Gy, once a day, 5 times/week.
  Interventions: Drug: TQB2450; Radiation: Intensity modulated radiotherapy

INTERVENTIONS:
Drug: TQB2450 — TQB2450 is a humanized monoclonal antibody targeting programmed death ligand-1 (PD-L1), which prevents PD-L1 from binding to PD-1 and B7.1 receptors on T cell surface, restores T cell activity, thus enhancing immune response and has potential to treat various types of tumors.
Radiation: Intensity modulated radiotherapy — Intensity-modulated conformal radiotherapy (IMRT) is a kind of three dimensional conformal radiotherapy, which requires the dose intensity in the radiation field to be adjusted according to certain requirements.

SUMMARY:
This is a study to evaluate the efficacy and safety of TQB2450 injection combination with Intensity-modulated Radiotherapy in patients with inoperable locally recurrent nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* 1. Understood and Signed an informed consent form; 2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1; Life expectancy ≥ 3 months; 3. Local recurrence of non-keratinizing nasopharyngeal carcinoma diagnosed by histopathology and/or cytology; Clinical stage: rT2-4N0-3M0 , RII-IVa phase (AJCC eighth edition); 4. The recurrence time is more than 12 months from the end of the first course of radiotherapy, without other systemic or local anti-tumor treatment; 5. At least one measurable lesion (based on RECIST 1.1); 6. Adequate laboratory indicators; 7. No pregnant or breastfeeding women, and a negative pregnancy test.

Exclusion Criteria:

* 1. Operable patients with local recurrence, including rT2 (the tumor is confined to the surface of the parapharyngeal space, and the distance from the internal carotid artery > 0.5 cm) and rT3 (the tumor is confined to the bottom wall of the sphenoid sinus, and the distance from the internal carotid artery and cavernous sinus > 0.5 cm) ; 2.Combined diseases and medical history:

  1. Accompanied by nasopharyngeal necrosis, radiation brain injury, severe neck fibrosis, or other ≥grade 3 radiation complications, the investigator has assessed that the risk is extremely high and not suitable for radiotherapy;
  2. Has other malignant tumors within 3 years;
  3. Unalleviated toxicity ≥ grade 1 due to any previous anticancer therapy;
  4. Has received major surgical treatment, open biopsy, or obvious traumatic injury within 28 days before the first administration;
  5. Long-term unhealed wounds or fractures;
  6. Arterial/venous thrombosis events occurred within 6 months, such as cerebrovascular accidents (including temporary ischemic attacks, cerebral; hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism;
  7. Has drug abuse history that unable to abstain from or mental disorders;
  8. Has any severe and/or uncontrollable disease. 3.Tumor-related symptoms and treatment:

  <!-- -->

  1. Diagnosed local recurrence and received surgery, chemotherapy, radiotherapy or other anti-cancer therapies before first administration;
  2. Has received NMPA approved Chinese patent medicines with anti-tumor indications;
  3. Has received relevant immunotherapy drugs for PD-1, PD-L1, CTLA-4, etc.;
  4. Uncontrollable pleural effusion, pericardial effusion or ascites that still needs to be drained repeatedly (as judged by the investigator); 4.Research and treatment related:

  <!-- -->

  1. Has vaccinated with vaccines or attenuated vaccines within 4 weeks prior to first administration;
  2. Have severe hypersensitivity after using monoclonal antibodies;
  3. Active autoimmune diseases that require systemic treatment (such as the use of disease-relieving drugs, corticosteroids, or immunosuppressive agents) occurred within 2 years before the start of the study treatment;
  4. Has immunodeficiency or received systemic glucocorticoid therapy or any other form of immunosuppressive therapy, and continue to use within 2 weeks of the first administration; 5.Has participated in other anti-tumor drug clinical trials within 4 weeks before the study; 6.According to the judgement of the investigators, there are other factors that may lead to the termination of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-04-29 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) | up to 48 weeks
  Percentage of participants achieving complete response (CR) and partial response (PR).

SECONDARY OUTCOMES:
Disease control rate（DCR） | up to 48 weeks
  Percentage of participants achieving complete response (CR) and partial response (PR) and stable disease (SD).
Duration of Response (DOR) | up to 48 weeks
  The time when the participants first achieved complete or partial remission to disease progression.
Progression-free survival (PFS) | up to 48 weeks
  PFS defined as the time from first dose until the first documented progressive disease (PD) or death from any cause.
12-month progression-free survival rate | up to 48 weeks
  12-month PFS defined as the time from first administration until the first documented progressive disease (PD) or death from any cause within 12 months.
12-month survival rate | up to 48 weeks
  12-month survival rate defined as the time from first administration to death from any cause within 12 months.
24-month survival rate | up to 96 weeks
  24-month survival rate defined as the time from first administration to death from any cause within 24 months.
Local regional recurrence-free survival (LRRFs) | up to 48 weeks
  The time interval between the patient's first medication and the appearance of local imaging progress.
Distant metastasis-free survival (DMFS) | up to 48 weeks
  The time interval between the patient's first medication and the appearance of distant metastasis imaging progression or death.
Overall survival (OS) | up to 96 weeks
  OS defined as the time from randomization to death from any cause. Participants who do not die at the end of the extended follow-up period, or were lost to follow-up during the study, were censored at the last date they were known to be alive.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Xia TL, Huang W, Liu YP, Feng ZK, Chen SY, Ding X, Peng L, Wu WB, Yu D, Yang AQ, Li X, Tang Y, He X, Hua YJ, You R, Chen MY. TQB2450 plus intensity-modulated radiotherapy in recurrent nasopharyngeal carcinoma: An open-label, single-arm, phase II trial. Med. 2025 Nov 14;6(11):100846. doi: 10.1016/j.medj.2025.100846. Epub 2025 Oct 8. PMID 41067232